CLINICAL TRIAL: NCT00167011
Title: Patterns of Coronary Artery Anatomy in Children With Congenital Heart Disease by Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9461700813
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Heart Diseases
Keywords: coronary artery
MeSH Terms: conditions — Heart Diseases

INTERVENTIONS:
Procedure: CT

SUMMARY:
To test the ability of electron beam CT in evalting the coronary artery pattern in children with congenital heart disease.

DETAILED DESCRIPTION:
To test the ability of electron beam CT in evalting the coronary artery pattern in children with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

- TOF, DORV, TGA, CCT

Exclusion Criteria:

-

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 1995-07; Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy

SECONDARY OUTCOMES:
sensitivity
specificity

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Jye Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan